CLINICAL TRIAL: NCT05428215
Title: Comparison of Pharmacokinetics of 17-Beta-Estradiol Via Oral Administration With Sublingual Placement Versus Oral Administration With Swallowing of 17-Beta-estradiol in Male-to-Female Transgender Patients
Brief Title: Comparison of PKs of 17-Beta-Estradiol Via Sublingual Placement Versus Swallowing in Male-to-Female Transgender Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to adequately recruit participants, need for additional study participants based on preliminary data collection
Sponsor: MaineHealth (Other)
Responsible Party: Principal Investigator, Katherine Davis, Physician- MH Obstetrics and Gynecology, MaineHealth
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1737257
Record Dates: First submitted 2022-01-11; First posted 2022-06-23 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Gender Dysphoria
Keywords: estradiol; gender-affirming estrogen
MeSH Terms: conditions — Gender Dysphoria | interventions — Estradiol

STUDY DESIGN:
Intervention Model Description: Each subject will take their individualized dose of 17B-estradiol tablet orally for 2 weeks and sublingually for 2 weeks. The subject will then take their same dose of 17B-estradiol via the other means of administration for 2 weeks. The order in which this occurs will be randomized.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PO then SL (Active Comparator): Subjects will administer 17-beta-estradiol orally (PO) for Study Day 1-14, followed by administration of 17-beta-estradiol sublingually (SL) for Study Day 15-28.
  Interventions: Drug: 17beta Estradiol
- SL then PO (Active Comparator): Subjects will administer 17-beta-estradiol sublingually (SL) for Study Day 1-14, followed by administration of 17-beta-estradiol orally (PO) for Study Day 15-28.
  Interventions: Drug: 17beta Estradiol

INTERVENTIONS:
Drug: 17beta Estradiol — Subjects will take individualized therapeutic dose of 17-beta-estradiol via sublingual and oral administration

SUMMARY:
This crossover study will investigate the pharmacokinetics of oral versus sublingual administration of 17-beta-estradiol in the trans-female population.

ELIGIBILITY:
Inclusion Criteria:

* English speaker
* Currently taking 17-beta-estradiol tablet daily via sublingual or oral route on dose therapeutic for gender-affirming therapy; steady dose for at least 4 weeks
* Serum estradiol and testosterone levels within target therapeutic range (75-200 pg/mL and <55 ng/dL, respectively)

Exclusion Criteria:

* Active or history of deep venous thrombosis/pulmonary embolism
* Active or recent (within the past year) arterial thromboembolic disease (e.g., stroke, myocardial infarction)
* Liver dysfunction
* History of breast cancer
* History of orchiectomy
* Known sensitivity or allergy to any components of the study medication
* Taking potent CYP3A4 inhibitors or inducers

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender male-to-female
Enrollment: 2 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Estradiol absorption | Over 24 hours
  Mean area under the curve of estradiol

SECONDARY OUTCOMES:
Peak serum estradiol | Peak over 24 hour period
  With subjects as own controls, compare peak E2 with sublingual vs oral administration
Serum estradiol Nadir | 24 hours from last estradiol administration
  Baseline serum estradiol level after 2 weeks of oral administration versus sublingual administration at same dose
Suppression of Testosterone | 24 hours from last estradiol administration on Study Day 14 and 28
  Testosterone level after 2 weeks of estradiol administration via oral and sublingual method, respectively
Serum estrone to estradiol ratio | Hours from administration of estradiol: 0, 1, 2, 4, 6, and 8 hours
  E1:E2 ratio over 24 hour period with sublingual vs oral administration
Sex hormone binding globulin | 0 hours from estradiol administration on Study Day 14 and 28
  SHBG after 2 weeks of estradiol sublingual vs oral administration

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Davis, MD, Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No